CLINICAL TRIAL: NCT04831554
Title: Comparison of the Efficacy of Single Tube Versus Multiple Tubes Drainage After Bullectomy and Pleurodesis for Primary Spontaneous Pneumothorax
Brief Title: Which is Better Between Single Chest Tube and Multiple Tubes Drainage in Primary Spontaneous Pneumothorax
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mashaohua1976-4
Record Dates: First submitted 2021-04-02; First posted 2021-04-05 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-04

CONDITIONS: Primary Spontaneous Pneumothorax
Keywords: number of chest tube; Bullectomy; Pleurodesis; Primary Spontaneous Pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single chest tube group (Experimental)
  Interventions: Procedure: single chest tube drainage
- multiple chest tubes group (No Intervention)

INTERVENTIONS:
Procedure: single chest tube drainage — place single chest tube after surgery of PSP
  Arms: single chest tube group

SUMMARY:
There was no evidence that the number of chest tube do effect to the recurrence of pneumothorax, which placed after thoracoscopic wedge resection together with mechanical pleurodesis.This study evaluates the efficacy of single chest tube versus multiple tubes drainage in spontaneous pneumothorax after VATS bullectomy and pleurodesis. After routine procedure the participants will randomized to either placed single chest tube or multiple chest tubes

DETAILED DESCRIPTION:
Primary spontaneous pneumothorax (PSP) occurs after the rupture of small bullae or a subpleural bleb in otherwise normal lungs. The indications for surgical treatment include persistent air leak after intercostal tube drainage, recurrent PSP, and contralateral PSP. The video-assisted thoracoscopic surgery (VATS) approach probably represents the treatment of choice for PSP.

The presence of a residual pleural space after surgery may be a factor associated with increased risk of recurrence. One possible hypothesis to explain the association between residual pleural space and recurrence of pneumothorax may be the failed pleurodesis due to lack of pleura-pleura apposition. Multiple chest tubes are effective in clinical practice, but there was no convinctive evidence that the number of chest tube do effect to the recurrence of pneumothorax, which placed after thoracoscopic wedge resection together with mechanical pleurodesis. This study evaluates the efficacy of single chest tube versus multiple tubes drainage in spontaneous pneumothorax after VATS bullectomy and pleurodesis.After routine procedure the participants will randomized to either placed multiple chest tubes or single chest tube.

The recurrence of the two group and other postoperative clinical parameters will be observed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by chest radiograph or CT as primary spontaneous pneumothorax
* Underwent bullectomy and pleurodesis
* Postoperative indwelling chest tubes

Exclusion Criteria:

* Secondary pneumothorax, traumatic pneumothorax and iatrogenic pneumothorax
* Previous surgery history
* People with severe comorbidities

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10-31 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
recurrence | 2 years after operation
  Recurrence of pneumothorax during 2 years follow-up

SECONDARY OUTCOMES:
complications | 30days after operation
  post-operation complications，such as air leakage

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiang L, Jiang G, Zhu Y, Hao W, Zhang L. Risk factors predisposing to prolonged air leak after video-assisted thoracoscopic surgery for spontaneous pneumothorax. Ann Thorac Surg. 2014 Mar;97(3):1008-13. doi: 10.1016/j.athoracsur.2013.10.031. Epub 2013 Dec 25. PMID 24370202
- [Background] Sudduth CL, Shinnick JK, Geng Z, McCracken CE, Clifton MS, Raval MV. Optimal surgical technique in spontaneous pneumothorax: a systematic review and meta-analysis. J Surg Res. 2017 Apr;210:32-46. doi: 10.1016/j.jss.2016.10.024. Epub 2016 Nov 3. PMID 28457339